CLINICAL TRIAL: NCT00931294
Title: Saliva Testosterone Increases in Choir Singer Beginners: a Randomised Controlled Trial to Test the Efficacy of Choir Singing in Irritable Bowel Syndrome (IBS) Patients
Brief Title: Saliva Testosterone Increases in Irritable Bowel Syndrome (IBS) Patients Beginning Choir Singing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stockholm University (Other)
Collaborators: The Swedish Research Council (Other Government); Region Stockholm (Other Government)
Responsible Party: Stress Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SI 5.1 2007-17
Record Dates: First submitted 2009-06-30; First posted 2009-07-02 (Estimated); Last update posted 2009-07-02 (Estimated); Status verified 2009-07

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Choir singing — Choir group participated in various relaxation, breathing and vocal exercises with the choir leader, and received the material "To Live with IBS" for home studies, weekly for 1 year. Saliva testosterone assessed 6 times per occasion; baseline, after 6, 9 and 12 months.
Behavioral: Information Group — Meet in groups, studying and discussing on the same materials under the direction of a group leader, weekly, for 1 year. Saliva testosterone assessed 6 times per occasion; baseline, after 6, 9 and 12 months.

SUMMARY:
The hypothesis was that a one-year experience of choir singing once a week is more beneficial than group discussions to saliva concentration of testosterone.

DETAILED DESCRIPTION:
The project aimed to study the health effects of regular choir singing for persons who are in a psychosomatic condition (Irritable Bowel syndrome - IBS). A group of IBS patients were randomized to choir singing or an information group were followed during one year with biological and psychosocial assessments. The choir group participated in various relaxation, breathing and vocal exercises with the choir leader, and received the material "To live with IBS" for home studies. At the same time a comparison group with IBS patients meet in groups, studying and discussing on the same materials under the direction of a group leader. Both groups meet once per week.

ELIGIBILITY:
Inclusion Criteria:

* IBS according to physician certificates.
* Wish to start choir singing but no such experience during past ten years.
* Acceptance of randomisation condition.

Exclusion Criteria:

* No serious somatic diseases.
* No abuse of alcohol or drugs.
* No ongoing acute psychiatric condition.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2006-05; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
More reduction in bowel pain according to standardised international IBS questionnaire in choir group than in study group after one year. | 1 year

SECONDARY OUTCOMES:
Significant increase in saliva testosterone concentration during study period in choir group. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Töres Theorell, MD, PhD, Professor, Principal Investigator — Stress Research Institute at Stockholm University
Locations (1):
- Stockholm, Sweden

REFERENCES:
- [Result] Christina Grape RN, Theorell T, Wikstrom BM, Ekman R. Choir singing and fibrinogen. VEGF, cholecystokinin and motilin in IBS patients. Med Hypotheses. 2009 Feb;72(2):223-5. doi: 10.1016/j.mehy.2008.09.019. Epub 2008 Oct 31. No abstract available. PMID 18951728
- See also: Stress Research Institute homepage — http://www.stressforskning.su.se